CLINICAL TRIAL: NCT05157594
Title: Pilot Study of hPG80 (Circulating Progastrin) as a Blood Biomarker for High-grade Glial Tumors
Brief Title: hPG80 (Circulating Progastrin) as a Blood Biomarker for High-grade Glial Tumors
Acronym: PROGLIO
Status: Completed | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Collaborators: ECS Progastrin (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-A01907-34
Record Dates: First submitted 2021-10-27; First posted 2021-12-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glial Cell Tumors
Keywords: Glial Cell Tumors; Progastrin; hPG80
MeSH Terms: conditions — Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: A fasting blood sample will be taken on the day of the beginning and the day of the end of the radiotherapy and during the adjuvant chemotherapy (every 3 cycles). A follow-up will be performed for 9 months, with a blood sample taken every three months on the day of the follow-up MRI.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Evaluation of plasma hPG80 concentrations by fasting blood samples. A total of seven 5 mL blood samples will be taken: Before radiation therapy; at the end of radiation therapy; at cycle 3 of chemotherapy; at cycle 6 of chemotherapy; 3 months after the end of treatment; 6 months after the end of treatment; and 9 months after the end of treatment.

SUMMARY:
PROGLIO is a French mono-centric study with longitudinal follow-up, in which patients with high grade brain tumors will be included. Blood samples will be taken during their therapeutic follow-up to evaluate plasma concentrations of hPG80 (circulating progastrin).

ELIGIBILITY:
Inclusion Criteria:

* Female or male 18 years of age or older.
* Patients with a high grade primary glial tumor (Astrocytoma grade 3; Glioblastoma; Anaplastic Oligodendroglioma)
* Patients scheduled to begin radiation and/or chemotherapy.
* Able to give informed consent to participate in the research.
* Enrolled in a social security plan or beneficiary of such a plan.

Exclusion Criteria:

* Patient under guardianship or curatorship
* Psychological disorder (cognitive disorders, vigilance disorders, etc.) or social reasons (deprivation of liberty by judicial or administrative decision) or geographical reasons that could compromise the medical follow-up of the trial.
* Refusal to participate.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female or male, 18 years of age or older, with a primary high-grade glial tumor (Astrocytoma Grade 3; Glioblastoma; Anaplastic Oligodendroglioma) who needs to initiate radiation and/or chemotherapy.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of hPG80 | From Radiotherapy 1st session to 9 month follow-up
  To evaluate plasma concentrations of hPG80 (circulating progastrin) during therapeutic and recurrence follow-up in patients with high-grade brain tumors.

SECONDARY OUTCOMES:
hPG80 concentration according to tumor progression | Through study completion, an average of 1 year and 6 months
  To study hPG80 concentration according to tumor progression in patients with high-grade brain tumor
Sensitivity of hPG80 concentration changes to irradiation | Through study completion, an average of 1 year and 6 months
  To evaluate the sensitivity of hPG80 concentration changes to irradiation in patients with high-grade brain tumor.
Interindividual variations of hPG80 concentration | Through study completion, an average of 1 year and 6 months
  To compare the plasma expression level of hPG80 in patients with high-grade brain tumor to study interindividual variations around and during disease management.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Pr, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casile M, Passildas J, Vire B, Molnar I, Durando X. hPG80 (circulating progastrin) as a blood biomarker for high-grade glial tumors: A pilot study. Front Neurol. 2023 Jan 11;13:1073476. doi: 10.3389/fneur.2022.1073476. eCollection 2022. PMID 36712425